CLINICAL TRIAL: NCT04397419
Title: Flying High - Exploring the Effect of Red Bull Energy Drink Intake After Autologous Microsurgical Breast Reconstruction
Brief Title: Red Bull Energy Drink Intake After Autologous Microsurgical Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Plastic Surgery Group AG by Prof. Jian Farhadi (Other)
Responsible Party: Principal Investigator, Dr. med. Nicole Speck, Prof. Dr. med. Jian Farhadi, Plastic Surgery Group AG by Prof. Jian Farhadi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-00493
Record Dates: First submitted 2020-05-17; First posted 2020-05-21 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 1 intervention group, 1 placebo group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group is administered a total of 750 ml Red Bull® Energy Drink at defined time-intervals.
  Interventions: Dietary Supplement: Red Bull Energy Drink
- Placebo group (Placebo Comparator): This group is administered a total of 750 ml still water at defined time-intervals.
  Interventions: Other: Still water

INTERVENTIONS:
Dietary Supplement: Red Bull Energy Drink — The intervention group receives 250 ml Red Bull Energy Drink 2-3 hours after surgery and 500 ml on postoperative day 1.
  Regimen:
  * 2-3 hours after surgery: 250 ml
  * Postoperative day 1: morning and noon (1-1-0-0) 250 ml
  Arms: Intervention group
Other: Still water — The control group receives 250 ml still water 2-3 hours after surgery and 500 ml on postoperative day 1.
  Regimen:
  * 2-3 hours after surgery: 250 ml
  * Postoperative day 1: morning and noon (1-1-0-0) 250 ml
  Arms: Placebo group

SUMMARY:
The success rate of autologous microsurgical breast reconstruction depends on adequate intraoperative and postoperative flap perfusion. Perfusion is optimized intraoperatively by a full hyperdynamic circulation and maintenance of a normal body temperature. Additional safe and simple postoperative measures to guarantee adequate perfusion pressure would be desirable. Recently, the effect of Red Bull® Energy Drink on cardiovascular and renal function, pain tolerance as well as performance has been studied in clinical trials involving healthy volunteers and athletes. Notably, an increase in blood pressure, heart rate, improved endothelial function and reduced pain perception have been observed. A better understanding of its effects in patients undergoing autologous microsurgical breast surgery would be of great value. When ingested in standard amounts, Red Bull® Energy Drink has been shown to be a safe beverage without notable side effects. The investigators prospectively study the effect of postoperative oral ingestion of Red Bull® Energy Drink on perfusion-related variables and patient recovery after autologous microsurgical breast reconstruction.

DETAILED DESCRIPTION:
All consecutive female patients receiving unilateral autologous microsurgical breast reconstruction starting from quarter I 2020 will be administered a total of either 750 ml Red Bull® Energy Drink (intervention group) or 750 ml still water (control group). The first dose of 250 ml Red Bull® Energy Drink or still water will be given 2-3 hours postoperatively. The following doses will be given on postoperative day 1 for breakfast (250 ml) and for lunch (250 ml).

The systolic and diastolic blood pressure as well as pulse will be measured non-invasively using a 24-hour ambulatory blood pressure monitor at regular intervals during the first postoperative 24 hours. Total fluid administered intraoperatively and postoperatively as well as intraoperative and postoperative administration of vasoactive drugs will be recorded. Daily urinary output will be measured during 24 hours after surgery. Pain levels will be measured on Numeric Rating Scale with values ranging from 0 to 10. Rate of operative re-explorations, flap loss and total length of primary hospital stay will be recorded. Wound healing and scarring will be assessed 1 month after surgery in our clinic and documented photographically.

The variables obtained from the intervention group receiving Red Bull® Energy Drink postoperatively will be compared with the corresponding variables of patients in the control group receiving the same amount of still water.

ELIGIBILITY:
Inclusion Criteria:

1. Indication: Patients undergoing unilateral autologous microsurgical breast reconstruction by Prof. Dr. med. Jian Farhadi, Dr. med. Alessia Lardi or Dr. med. Doris Babst
2. Female participants ≥ 18 and ≤ 70 years of age
3. Able to give written informed consent prior to participation in the study, which includes ability to comply with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. History of arterial hypertension*
2. History of cardiac rhythm disorder*
3. History of Diabetes mellitus*
4. History of gastric or duodenal ulcer*
5. History of hyperthyroidism or hypothyroidism*
6. Current use of antihypertensive drugs, antiarrhythmic drugs, thyroid hormones (e.g. Euthyrox)*
7. Allergy or intolerance to component of Red Bull® Energy Drink
8. Not fulfilling inclusion criteria. * as diagnosed by the GP in the referral letter

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Until 2 hours after last drink ingestion
  Difference in mean systolic blood pressure [mmHg] between the intervention group and the control group at 15/30/45/60/75/90/105/120min after each of 3 Red Bull (intervention group)/water (control group) applications

CONTACTS AND LOCATIONS:
Overall Officials: Jian Farhadi, M.D., Prof., Principal Investigator — University of Basel, Plastic Surgery Group AG by Prof. Jian Farhadi, Switzerland
Locations (1):
- Klinik Pyramide am See, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Speck NE, Michalak M, Dreier K, Babst D, Lardi AM, Farhadi J. Effect of the Red Bull Energy Drink on Perfusion-Related Variables in Women Undergoing Microsurgical Breast Reconstruction: Protocol and Analysis Plan for a Prospective, Multicenter Randomized Controlled Trial. JMIR Res Protoc. 2023 May 9;12:e38487. doi: 10.2196/38487. PMID 37159251